CLINICAL TRIAL: NCT06466473
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE-DOSE, 2-WAY CROSSOVER, PIVOTAL BIOEQUIVALENCE STUDY COMPARING 50-MG CHEWABLE DILANTIN® INFATABS® MANUFACTURED AT VEGA BAJA (PUERTO RICO) AND ASCOLI (ITALY) IN HEALTHY ADULT PARTICIPANTS UNDER FASTING CONDITIONS
Brief Title: A Study to Learn How Different Forms of The Study Medicine Called Phenytoin Are Taken up Into the Blood in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: A4121018
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: Bioequivalence; Phenytoin; Healthy participants; Pharmacokinetic; Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phenytoin manufactured at Vega Baja site (Active Comparator)
  Interventions: Drug: Phenytoin (Vega Baja)
- Phenytoin manufactored at Ascoli site (Experimental)
  Interventions: Drug: Phenytoin (Ascoli)

INTERVENTIONS:
Drug: Phenytoin (Ascoli) — Phenytoin 50mg chewable tablets
  Arms: Phenytoin manufactored at Ascoli site
Drug: Phenytoin (Vega Baja) — Phenytoin 50mg chewable tablets
  Arms: Phenytoin manufactured at Vega Baja site

SUMMARY:
The purpose of this study is to understand how the different formulation of phenytoin is taken up into the blood in Healthy Adults.

This study is seeking healthy adult participants. All the study participants will receive Phenytoin 50 mg chewable tablets manufactured at Ascoli and Vega Baja manufacturing site.

We will measure how the phenytoin will be taken up into the blood in Healthy Adults following oral dosing of Phenytoin.

This will help us determine if the Phenytoin 50 mg chewable tablets manufactured at Ascoli and Vega Baja manufacturing site are similar or not.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male participants and female participants of non-childbearing potential aged 18 years or older determined by medical evaluation including detailed medical history, complete physical examination, blood pressure (BP) and pulse rate measurement, 12-lead electrocardiogram (ECG), and/or clinical laboratory tests.
2. Body mass index (BMI) of 16-32 kg/m2; and a total body weight >45 kg (100 lb).

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Female participants of childbearing potential; pregnant female participants; breastfeeding female participants; male participants with partners currently pregnant; male participants able to father children who, with their partner(s) are at risk for pregnancy and are unwilling or unable to use a highly effective method of contraception.
3. History of hypersensitivity to phenytoin or its inactive ingredients.
4. Any medical or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
5. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days prior to the first dose of study intervention.
6. Current use of any prohibited concomitant medication(s).
7. History of febrile illness within 5 days prior to first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Profile From Time Zero to the Time of Last Quantifiable Concentration (AUClast) | 72 hours
Maximum Observed Plasma Concentration (Cmax) of Phenytoin | 72 hours

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) According to Seriousness | Baseline, up to 35 days post last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A4121018